CLINICAL TRIAL: NCT03130322
Title: Neurophysiological Correlates of Sleep Motor Consolidation Following Motor Imagery Practice
Brief Title: SLeep and IMagery Correlates (SOMMEIL-IMAGERIE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0676
Record Dates: First submitted 2017-03-10; First posted 2017-04-26 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- NightPP (Experimental): Participants of the NightPP will be subjected to one MRI session and two MEG recording sessions: the first one before a physical practice session of the two motor tasks investigated in the study, and second MEG session right after practice.
  Interventions: Other: Imagery and Sleep questionnaires; Other: MEG recordings (pre-test); Other: Practice session; Other: MEG recordings (Post-test); Other: MRI
- NightMI (Experimental): Participants of the NightMI will be subjected to one MRI session and two MEG recording sessions: the first one before a motor imagery practice session of the two motor tasks investigated in the study, and second MEG session right after practice.
  Interventions: Other: Imagery and Sleep questionnaires; Other: MEG recordings (pre-test); Other: Practice session; Other: MEG recordings (Post-test); Other: MRI
- NightCtrl (Experimental): Participants of the NightCtrl will be subjected to one MRI session and two MEG recording sessions: the first one before a mental rotation practice session, a second MEG session right after practice,and second MEG session right after practice.
  Interventions: Other: Imagery and Sleep questionnaires; Other: MEG recordings (pre-test); Other: Practice session; Other: MEG recordings (Post-test); Other: MRI
- Day (Experimental): Participants of the NightMI will be subjected to one MRI session and two MEG recording sessions: the first one before a motor imagery practice session of the two motor tasks investigated in the study, and second MEG session right after practice.
  Interventions: Other: Imagery and Sleep questionnaires; Other: MEG recordings (pre-test); Other: Practice session; Other: MEG recordings (Post-test); Other: MRI

INTERVENTIONS:
Other: Imagery and Sleep questionnaires — Participants complete a motor imagery questionnaire to assess their ability to form vivid mental images, as well as sleep questionnaires to control the quality of their sleep
Other: MEG recordings (pre-test) — Participants of the Day group perform two motor tasks (a finger sequential motor task and an adaptation motor task using a trackball) in the MEG, during a pre-test (Day 1 - 9h).
  Task 1: Participants perform an 8-digit motor sequential task where each finger (except the thumb) is used twice. Performance is assessed by using a 4-keys keyboard. Participants are required to keep their fingers on the keys to minimize amplitude are instructed to tap the sequence as few errors as possible Task 2: Participants perform a motor adaptation task requiring scrolling a trackball to superimpose a geometric shape on another one, strictly similar but presented from another angle, as fast as possible.
Other: Practice session — Participants of the Day group perform a block of motor imagery practice of the two motor tasks.
Other: MEG recordings (Post-test) — Participants perform the two motor tasks in the MEG (post-test, strictly similar to the pre-test)
Other: MRI — The registration of the brain anatomy of each participant will be done by MRI 3D / T the week before the first experimental session.

SUMMARY:
This study is designed to determine the neural networks underlying the sleep-related motor consolidation process following motor imagery practice. While beneficial effects of sleep are expected for sequential movement but not for adaptation motor tasks, the corresponding neuroanatomical correlates have not yet been investigated when participants acquired the motor tasks through mental practice. Data should substantially promote how designing motor imagery interventions targeting (re)learning and/or motor recovery in patients suffering from motor disorders.

ELIGIBILITY:
Inclusion Criteria:

* Healthy right-handed persons without neurologic disease
* Persons having signed informed consent for a neuroimagery study

Exclusion Criteria:

* Persons under curatorship or any administrative/judicial measure
* Participants refusing to be informed of the results of the experiment
* Pregnant women
* Participants with contraindications to the MEG examination: head size, presence of a neurostimulator, steel pivot for the root canal, metallic fragments, ear implants, metal screws in the body or mouth.
* Persons using a pacemaker, insulin pump, or working regularly with iron filings
* Claustrophobic persons

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2017-12-09 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Evidence of MEG correlates of sleep motor consolidation (day 1) | Day 1 at 19h00 [post-training] (Groups 1, 2 and 3) OR Day 1 at 9h00 [post-training] (Group 4)
  The investigator will use Single Aperture Magnetometry, i.e. a minimum variance beamformer mapping the spatial distribution of event-related desynchronizations and synchronizations within a predetermined frequency domain (Beta oscillations 15-35 Hz). The time course of MEG Beta power will be considered, and Granger causal connectivity analyses will be performed to investigate relationships between cortical motor regions.
Evidence of MEG correlates of sleep motor consolidation (day 2) | Day 2 at 9h00 [Retention test] (Groups 1, 2 and 3) OR Day 1 at 19h00 [Retention test] (Group 4)
  The investigator will use Single Aperture Magnetometry, i.e. a minimum variance beamformer mapping the spatial distribution of event-related desynchronizations and synchronizations within a predetermined frequency domain (Beta oscillations 15-35 Hz). The time course of MEG Beta power will be considered, and Granger causal connectivity analyses will be performed to investigate relationships between cortical motor regions.

SECONDARY OUTCOMES:
Time needed to complete the motor tasks (day 1) | Day 1 at 19h00 [post-training] (Groups 1, 2 and 3) OR Day 1 at 9h00 [post-training] (Group 4)
  The investigators will measure the time needed to complete the motor tasks needed to complete each motor task (finger sequential tasks OR motor adaptation task).
Evidence of MEG correlates of sleep motor consolidation | Day 2 at 9h00 [Retention test] (Groups 1, 2 and 3) OR Day 1 at 19h00 [Retention test] (Group 4)
  The investigators will use Single Aperture Magnetometry, i.e. a minimum variance beamformer mapping the spatial distribution of event-related desynchronizations and synchronizations within a predetermined frequency domain (Beta oscillations 15-35 Hz). The time course of MEG Beta power will be considered, and Granger causal connectivity analyses will be performed to investigate relationships between cortical motor regions.
Accuracy of the motor tasks | Day 1 at 19h00 [post-training] (Groups 1, 2 and 3) OR Day 1 at 9h00 [post-training] (Group 4)
  The investigators will measure the number of errors and correct trials for each motor task (finger sequential tasks OR motor adaptation task).
Time needed to complete the motor tasks | Day 2 at 9h00 [Retention test] (Groups 1, 2 and 3) OR Day 1 at 19h00 [Retention test] (Group 4)
  The investigators will measure the time needed to complete each motor task (finger sequential tasks OR motor adaptation task).
Accuracy of the motor tasks 2 | Day 2 at 9h00 [Retention test] (Groups 1, 2 and 3) OR Day 1 at 19h00 [Retention test] (Group 4)
  The investigators will measure the number of errors and correct trials for each motor task (finger sequential tasks OR motor adaptation task).

CONTACTS AND LOCATIONS:
Overall Officials: Alain Nicolas, MD, Principal Investigator — CH le Vinatier
Locations (1):
- CH le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Rienzo F, Debarnot U, Daligault S, Delpuech C, Doyon J, Guillot A. Brain plasticity underlying sleep-dependent motor consolidation after motor imagery. Cereb Cortex. 2023 Nov 27;33(23):11431-11445. doi: 10.1093/cercor/bhad379. PMID 37814365